CLINICAL TRIAL: NCT02943473
Title: A Phase 2 Study of the Effect of the Bruton's Tyrosine Kinase Inhibitor Ibrutinib on Disease Response in Patients With High Risk Smoldering Multiple Myeloma
Brief Title: Study on the Effect of Ibrutinib on High Risk Smoldering Multiple Myeloma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual and risk/benefit ratio.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Principal Investigator, Ajai Chari, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1867
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: High Risk Smoldering Multiple Myeloma
Keywords: Smoldering multiple myeloma; myeloma; smoldering; ibrutinib
MeSH Terms: conditions — Smoldering Multiple Myeloma; Neoplasms, Plasma Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Ibrutinib (trademark name is IMBRUVICA®). 560 mg dose administered on a continuous basis
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib is a type of drug called a "kinase inhibitor." Kinases are proteins inside cells that help cells live and grow. Ibrutinib blocks a specific kinase protein in our bodies. This protein is thought to be very important in helping blood cancer cells live and grow. By blocking this kinase protein, ibrutinib stops cancer cells from growing.
  Other Names: IMBRUVICA

SUMMARY:
The purpose of this research study is to test whether the drug ibrutinib (trademark name: IMBRUVICA®) is effective at preventing the development of multiple myeloma in people who currently have smoldering myeloma. The researchers conducting this trial) have reason to believe that ibrutinib can delay the development of multiple myeloma, thus giving people who currently have smoldering myeloma a longer period of time when they feel healthy and well.

Smoldering myeloma is an abnormal condition that is considered to be an early phase of the disease multiple myeloma. In this disorder, there is an abnormal growth of plasma cells, which is a type of blood cell found in the bone marrow. This growth is not as severe in people with smoldering myeloma as it is in multiple myeloma, so people with smoldering myeloma do not have any symptoms and tend to feel well. However, they have a higher risk of developing multiple myeloma than people in the general population.

Some people with smoldering myeloma are at an especially high risk of developing myeloma - 50% of these people will develop multiple myeloma 2 years after they are diagnosed with smoldering myeloma. The investigators identify these people by looking at the amount of myeloma in the bone marrow (called "bone marrow plasma cell percentage") and the amount of myeloma protein (called "serum protein electrophoresis" and "serum free light chain assay") in the blood. To be considered high risk, individuals must have highly abnormal levels for these tests.

Based upon current guidelines, people with smoldering myeloma do not require any treatment. However, known is that many of these people will develop multiple myeloma in the near future. Currently there have been no proven and effective way of preventing these people from developing multiple myeloma, which remains an incurable disease.

DETAILED DESCRIPTION:
This is a phase 2, open-label, single center, prospective pilot study designed to assess the efficacy of ibrutinib in subjects with high risk smoldering multiple myeloma.

All enrolled subjects will be treated with ibrutinib 560 mg (4 capsules, each containing 140 mg) taken PO daily for 12 cycles (28 days each). If a subject demonstrates benefit from ibrutinib, therapy may be extended beyond 12 cycles to a maximum of 2 years. Subjects who progress and meet criteria for symptomatic multiple myeloma will be withdrawn from study.

An initial cohort of 15 subjects will be accrued. If 4 or more patients progress to symptomatic myeloma in one year, then the study will be reviewed with the FDA to determine whether to employ a higher dose of ibrutinib, or to stop for futility. Otherwise, 21 additional patients will be accrued for a total sample size of 36.

ELIGIBILITY:
Inclusion Criteria Disease Related

1. High risk SMM, defined as follows by Mayo Clinic criteria:

   1. Bone marrow plasma cells between 10% and 60%
   2. Serum M-protein ≥ 3 g/dL [except IgA ≥ 2 g/dL] or urine M-protein > 500 mg per 24 hours
   3. Serum free light chain ratio < 0.126 or > 8; an involved to uninvolved ratio of ≥ 100 is permitted
   4. Measurable disease, defined as: M-protein ≥ 1 g/dL OR Bence-Jones protein (BJP) > 200 mg/24 hr OR involved free light chain > 100 mg/dL
2. Diagnosed with SMM within the last 4 years

Laboratory

1. Adequate hematologic function independent of transfusion and growth factor support for at least 7 days prior to screening, with the exception of pegylated G-CSF (pegfilgrastim) and darbopoetin which require at least 14 days prior to screening defined as:

   * Absolute neutrophil count > 750 cells/mm3 (1.0 x 109/L).
   * Platelet count > 75,000 cells/mm3 (75 x 109/L).
2. Adequate hepatic and renal function defined as:

   * Serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN).
   * Estimated creatinine clearance ≥ 30 ml/min (Cockcroft-Gault)
   * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin, in which case the total bilirubin should be < 3 x ULN)
3. PT/INR < 1.5 x ULN and PTT (aPTT) < 1.5 x ULN

   Demographic
4. Men and women ≥ 18 years of age
5. Eastern Cooperative Oncology Group (ECOG) performance status of < 2

Exclusion Criteria Disease-Related

1. No end organ damage attributable to a plasma cell disorder, defined as having ANY of the following:

   1. Hypercalcemia: Serum calcium > 1 mg/dL above the upper limit of normal or > 11 mg/dL
   2. Renal insufficiency: Serum creatinine > 2 mg/dL or creatinine clearance < 30 mL per min
   3. Anemia: Hemoglobin value > 2 g/dL below the upper limit of normal or a hemoglobin value < 10 g/dL
   4. Bone lesions: One or more lytic lesions on skeletal radiography, CT, MRI, PET-CT, or PET-MRI
2. Bone marrow plasma cells < 10% or > 60%
3. Has received prior anti-myeloma therapy of any type
4. Has received prior bisphosphonate therapy
5. Has received an investigational drug, investigational vaccine, or has used an investigational medical device within 4 weeks or 4 half-lives, whichever is longer, before Cycle 1, Day 1 of study therapy
6. Osteoporosis, defined as having a T-score on DEXA of ≤ -2.5

Concurrent Conditions

1. History of other malignancies, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
2. Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc). Any use of corticosteroids EITHER for > 14 days OR at dosages > 20 mg/day of prednisone or equivalent is prohibited.
3. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
4. Recent infection requiring systemic treatment that was completed ≤ 14 days before the first dose of study drug
5. Known bleeding disorders (eg, von Willebrand's disease) or hemophilia
6. History of stroke or intracranial hemorrhage within 6 months prior to enrollment
7. Known HIV, HCV or HBV infection. Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
8. Any uncontrolled active systemic infection
9. Major surgery within 4 weeks of first dose of study drug
10. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigators' opinion, could compromise the subject's safety or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Chari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from May 2017 through June 2019
Groups:
- Ibrutinib: Ibrutinib (trademark name is IMBRUVICA®). 560 mg dose taken PO daily for 12 cycles (28 days each).
  Ibrutinib: Ibrutinib is a type of drug called a "kinase inhibitor." Kinases are proteins inside cells that help cells live and grow. Ibrutinib blocks a specific kinase protein in our bodies. This protein is thought to be very important in helping blood cancer cells live and grow. By blocking this kinase protein, ibrutinib stops cancer cells from growing.
Period: Overall Study
Arm/Group | Ibrutinib
Started | 9
Completed | 3
Not Completed | 6
Not completed — enrolled but not dosed | 1
Not completed — screen failure | 1
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 3
  60 years and older | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Without Symptomatic Myeloma
Description: Disease response - the proportion of patients with high risk smoldering multiple myeloma who do not progress to symptomatic myeloma as defined by the IMWG.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 7
Participants | 5

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate, defined as partial response or better per IMWG criteria. (IMWG response criteria are - Complete Response, Very good partial response, partial response, Minimal response, stable disease, and progressive disease)
Time Frame: up to 1 year
Reporting Status: Not Posted, anticipated posting 2021-03

3. Secondary Outcome: Bone Density Changes
Description: Changes in bone density, particularly in patients with osteopenia (defined as T-score on bone densitometry testing (DEXA) of -1 to -2.5).
Time Frame: baseline and one year
Reporting Status: Not Posted, anticipated posting 2021-03

4. Secondary Outcome: PET-MRI Changes
Description: Changes in PET-MRI, particularly in patients with osteopenia
Time Frame: baseline and one year
Reporting Status: Not Posted, anticipated posting 2021-03

5. Secondary Outcome: Change in Serum Interleukin-6 (IL-6)
Description: Bone Related Biomarker Changes
Time Frame: baseline and up to one year
Reporting Status: Not Posted, anticipated posting 2021-03

6. Secondary Outcome: Change in Serum Stromal Cell-derived Factor-1 (SDF-1)
Description: Bone Related Biomarker Changes
Time Frame: baseline and up to one year
Reporting Status: Not Posted, anticipated posting 2021-03

7. Secondary Outcome: Change in Serum Receptor Activator of Nuclear-factor Kappa B Ligand (RANKL)
Description: Bone Related Biomarker Changes
Time Frame: baseline and up to one year
Reporting Status: Not Posted, anticipated posting 2021-03

8. Secondary Outcome: Change in Serum Macrophage Inflammatory Protein-1α (MIP-1α)
Description: Bone Related Biomarker Changes
Time Frame: baseline and up to one year
Reporting Status: Not Posted, anticipated posting 2021-03

9. Secondary Outcome: Change in Serum Dickkopf-1 (DKK-1)
Description: Bone Related Biomarker Changes
Time Frame: baseline and up to one year
Reporting Status: Not Posted, anticipated posting 2021-03

10. Secondary Outcome: Change in Serum C-terminal Telopeptide (CTX)
Description: Bone Related Biomarker Changes
Time Frame: baseline and up to one year
Reporting Status: Not Posted, anticipated posting 2021-03

11. Secondary Outcome: Change in Urine N-terminal Telopeptide (NTx)
Description: Bone Related Biomarker Changes
Time Frame: baseline and up to one year
Reporting Status: Not Posted, anticipated posting 2021-03

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=3)
Headache (General disorders) | 1 (1)
Tingling in Tongue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Irregular menses (Reproductive system and breast disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Loose stools (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Left musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Elevated AST (Hepatobiliary disorders) | 1 (1)
Elevated ALT (Investigations) | 1 (2)
Blateral ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee discomfort right (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Metabolism and nutrition disorders) | 1 (1)
Groin pain right (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT02943473/Prot_SAP_000.pdf